CLINICAL TRIAL: NCT02557646
Title: An Observational Study to Assess the Effect of Cumulative Ribavirin Dose in Participants With Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22453
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pegasys + Copegus: Treatment naive participants with confirmed chronic hepatitis C who are started on combined Pegasys-Copegus treatment in accordance with current guidelines and SPCs, and whose treatment has been approved by the Interferon Committee.
  Interventions: Biological: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Biological: Peginterferon alfa-2a — Participants received pegylated interferon subcutaneous injection in accordance with current guidelines and SPCs.P
  Other Names: Pegasys
Drug: Ribavirin — Participants received ribavirin 200 mg film-coated tablet in accordance with current guidelines and SPCs.
  Other Names: Copegus

SUMMARY:
The purpose of this open-label, non-randomized, single-arm, multicentre observational study is to investigate the influence of the cumulative dose (total administered dose/ planned dose) of ribavirin on the sustained virologic response (SVR) in participants who have been receiving combination therapy with pegylated interferon alfa-2a (Pegasys) and ribavirin (Copegus).

ELIGIBILITY:
Inclusion Criteria:

* Participants with serologically confirmed chronic hepatitis C
* Participants using and accepting a double method of contraception

Exclusion Criteria:

* Participants not approved by the national treatment guideline or the Interferon Committee for combined pegylated interferon-ribavirin treatment
* Contraindications in the summary of product characteristics of pegylated interferon alpha-2a and ribavirin
* Participants previously treated with pegylated interferon and/or ribavirin
* Hepatitis B and Human Immunodeficiency Virus co-infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment naive participants with confirmed chronic hepatitis C who are started on combined Pegasys-Copegus treatment in accordance with current guidelines and SPCs, and whose treatment has been approved by the Interferon Committee.
Sampling Method: Non-Probability Sample
Enrollment: 697 (Actual)
Dates: Start 2009-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Hungary (20):
  - Ajka
  - Balassagyarmat
  - Békéscsaba
  - Budapest
  - Debrecen
  - Győr
  - Gyula
  - Kaposvár
  - Kecskemét
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Sopron
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Tatabánya
  - Zalaegerszeg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 697 participants enrolled in the study, only 693 participants provided evaluable data. One participant did not receive peginterferon alfa-2a/ribavirin combination therapy, while 3 participants received combination therapy only for a very short time.
Groups:
- Peginterferon Alfa-2a + Ribavirin: Treatment naive participants with confirmed chronic hepatitis C who started combination therapy with peginterferon alfa 2a (Pegasys) and ribavirin (Copegus) in accordance with current guidelines and summary of product characteristics, upon decision of the treating physician, considering each participant's individual response, received combination therapy for 24, 48 or 72 weeks, followed by a 24-week follow-up period.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Started | 693
Completed | 417
Not Completed | 276
Not completed — Adverse Event | 40
Not completed — Death | 1
Not completed — Lack of Efficacy | 186
Not completed — Withdrawal by Subject | 18
Not completed — Lost to Follow-up | 17
Not completed — Other | 14

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all enrolled participants who provided evaluable data for the study.
Groups:
- Peginterferon Alfa-2a + Ribavirin: Treatment naive participants with confirmed chronic hepatitis C who started combination therapy with peginterferon alfa 2a and ribavirin in accordance with current guidelines and summary of product characteristics, upon decision of the treating physician, considering each participant's individual response, received combination therapy for 24, 48 or 72 weeks, followed by a 24-week follow-up period.
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 693
Age, Continuous [Mean (Standard Deviation); unit: years] — Out of total 693 participants in ITT population, data for only 692 participants was available for this baseline measure.
  years | 50.35 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 382
  Male | 311

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response (SVR) According to Cumulative Dose of Ribavirin
Description: Determination of hepatitis C virus (HCV) titers was performed using COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C, at Weeks 4, 12 and 24 of the treatment period (and, optionally, at the end of treatment [EOT] visit), and at the end of the 24-week follow-up period. Negative HCV titers measured at Weeks 4, 12, 24, and at EOT were interpreted as virological response, and negative HCV titers measured at the end of the 24-week follow-up period were interpreted as SVR. Percentage of participants achieving SVR in each cumulative dose group is presented. Cumulative dose was calculated as: (administered dose divided by planned dose) multiplied by 100.
Time Frame: 24 weeks after EOT (maximum up to 96 Weeks)
Population: ITT Population. Here, 'N' (number of participants analyzed) signifies the number of participants analyzed for this outcome measure and 'n' signifies the number of participants analyzed for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 406
percentage of participants
  Cumulative dose of ribavirin <60% (n=35) | 54.29
  Cumulative dose of ribavirin = 60-69% (n=23) | 60.87
  Cumulative dose of ribavirin = 70-79% (n=32) | 53.13
  Cumulative dose of ribavirin = 80-89% (n=52) | 50.00
  Cumulative dose of ribavirin >90% (n=264) | 68.56
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin; Cumulative dose of ribavirin >90%: the relationship between cumulative dose and SVR response in participants in whom the cumulative dose of ribavirin exceeded 90% was analyzed using Chi-square test; Test type: Superiority or Other; p = 0.0437, Chi-squared

2. Secondary Outcome: Percentage of Participants With Virologic Response
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. Negative HCV titers measured at Weeks 4, 12, 24 and at EOT were interpreted as virological response.
Time Frame: Week 4, 12, 24 and at EOT (maximum up to 72 weeks)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 693
percentage of participants
  Week 4 | 18.7
  Week 12 | 32.7
  Week 24 | 14.8
  EOT | 1.8

3. Secondary Outcome: Percentage of Participants With Virologic Response According to Starting Dose of Ribavirin
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. Negative HCV titers measured at Weeks 4, 12, 24 and at EOT were interpreted as virological response. Percentage of participants achieving virological response in each dose group is presented.
Time Frame: Up to EOT (maximum up to 72 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 690
percentage of participants
  Starting dose of ribavirin = 200mg (n=1) | 0.00
  Starting dose of ribavirin = 400mg (n=2) | 50.00
  Starting dose of ribavirin = 600mg (n=3) | 66.67
  Starting dose of ribavirin = 800mg (n=35) | 77.14
  Starting dose of ribavirin = 1000mg (n=277) | 67.15
  Starting dose of ribavirin = 1200mg (n=332) | 68.67
  Starting dose of ribavirin = 1400mg (n=40) | 67.50
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin; The relationship between the starting dose ribavirin and virological response was analyzed using Chi-square test; Test type: Superiority or Other; p = 0.6859, Chi-squared

4. Secondary Outcome: Percentage of Participants With SVR According to Starting Dose of Ribavirin
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. Negative HCV titers measured at Weeks 4, 12, 24, and at EOT were interpreted as virological response, and negative HCV titers measured at the end of the 24-week follow-up period were interpreted as SVR. Percentage of participants achieving SVR in each dose group is presented.
Time Frame: 24 weeks after EOT (maximum up to 96 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 660
percentage of participants
  Starting dose of ribavirin = 200mg (n=1) | 0.00
  Starting dose of ribavirin = 400mg (n=1) | 0.00
  Starting dose of ribavirin = 600mg (n=3) | 66.67
  Starting dose of ribavirin = 800mg (n=33) | 60.61
  Starting dose of ribavirin = 1000mg (n=262) | 43.13
  Starting dose of ribavirin = 1200mg (n=321) | 44.86
  Starting dose of ribavirin = 1400mg (n=39) | 38.46
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin; The relationship between the starting dose ribavirin and sustained virological response (SVR) was analyzed using Chi-square test; Test type: Superiority or Other; p = 0.3740, Chi-squared

5. Secondary Outcome: Percentage of Participants With Virologic Response According to Body Weight-normalized Dose of Ribavirin
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. Negative HCV titers measured at Weeks 4, 12, 24, and at EOT were interpreted as virological response. Percentage of participants achieving virological response in each body weight-normalized (measured in milligram per kilogram per day [mg/kg/day]) dose group is presented.
Time Frame: Up to EOT (maximum up to 72 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 691
percentage of participants
  Ribavirin dose <5mg/kg/day (n=5) | 40.00
  Ribavirin dose = 5-10 mg/kg/day (n=33) | 90.91
  Ribavirin dose = 10-15 mg/kg/day (n=383) | 68.93
  Ribavirin dose = 15-20 mg/kg/day (n=251) | 64.94
  Ribavirin dose >20mg/kg/day (n=19) | 68.42
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin; The relationship between the body weight-normalized dose of ribavirin and virological response was analyzed using Chi-square test; Test type: Superiority or Other; p = 0.0263, Chi-squared, Corrected

6. Secondary Outcome: Percentage of Participants With SVR According to Body Weight-normalized Dose of Ribavirin
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. Negative HCV titers measured at Weeks 4, 12, 24, and at EOT were interpreted as virological response, and negative HCV titers measured at the end of the 24-week follow-up period were interpreted as SVR. Percentage of participants achieving SVR in each body weight-normalized dose group is presented.
Time Frame: 24 weeks after EOT (maximum up to 96 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 661
percentage of participants
  Ribavirin dose <5mg/kg/day (n=5) | 0.00
  Ribavirin dose = 5-10 mg/kg/day (n=31) | 54.84
  Ribavirin dose = 10-15 mg/kg/day (n=368) | 41.03
  Ribavirin dose = 15-20 mg/kg/day (n=239) | 48.54
  Ribavirin dose >20mg/kg/day (n=18) | 55.56
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin; The relationship between the body weight-normalized dose of ribavirin and sustained virological (SVR) response was analyzed using Chi-square test; Test type: Superiority or Other; p = 0.0475, Chi-squared

7. Secondary Outcome: Percentage of Participants With Virologic Response According to Dose Reduction of Ribavirin
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. Negative HCV titers measured at Weeks 4, 12, 24, and at EOT were interpreted as virological response. Percentage of participants achieving virological response in each dose-reduction group (none, dose reduction within 12 weeks, dose reduction after 12 weeks, dose reduction not specified) is presented.
Time Frame: Up to EOT (maximum up to 72 weeks)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 693
percentage of participants
  None (n=443) | 67.49
  Within 12 weeks (n = 140) | 65.71
  After 12 weeks (n = 78) | 79.49
  Not Specified (n =32) | 62.50

8. Secondary Outcome: Percentage of Participants With SVR According to Dose Reduction of Ribavirin
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. Negative HCV titers measured at Weeks 4, 12, 24 and at EOT were interpreted as virological response, and negative HCV titers measured at the end of the 24-week follow-up period were interpreted as SVR. Percentage of participants achieving SVR in each dose-reduction group (none, dose reduction within 12 weeks, dose reduction after 12 weeks, dose reduction not specified) is presented.
Time Frame: 24 weeks after EOT (maximum up to 96 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 443
percentage of participants
  None (n=280) | 70.00
  Within 12 weeks (n = 87) | 57.47
  After 12 weeks (n = 57) | 63.16
  Not Specified (n =19) | 68.42

9. Secondary Outcome: Percentage of Participants With Virologic Response According to Interleukin-28B (IL-28B) Polymorphism
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. Negative HCV titers measured at Weeks 4, 12, 24 and at EOT were interpreted as virological response. Percentage of participants achieving virological response for each IL-28B allele (CC allele, CT allele, TT allele) is presented.
Time Frame: Up to EOT (maximum up to 72 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 97
percentage of participants
  CC Allele (n = 26) | 84.62
  CT Allele (n = 52) | 65.38
  TT Allele (n = 19) | 73.68

10. Secondary Outcome: Percentage of Participants With SVR According to IL-28B Polymorphism
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. Negative HCV titers measured at Weeks 4, 12, 24 and at EOT were interpreted as virological response, and negative HCV titers measured at the end of the 24-week follow-up period were interpreted as SVR. Percentage of participants achieving SVR for each IL-28B allele (CC allele, CT allele, TT allele) is presented.
Time Frame: 24 weeks after EOT (maximum up to 96 Weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 94
percentage of participants
  CC Allele (n = 25) | 64.00
  CT Allele (n = 51) | 39.22
  TT Allele (n = 18) | 33.33

11. Secondary Outcome: Percentage of Participants With Viral Relapse or Breakthrough
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. In participants with virological response, positive HCV titers measured during 24-week follow-up was interpreted as viral relapse, and positive HCV titers measured during the treatment period was interpreted as viral breakthrough. Percentage of participants with no relapse/breakthrough (none), with relapse, and with breakthrough is reported.
Time Frame: Up to 24 weeks after EOT (maximum up to 96 weeks)
Population: ITT Population showing virological response. Here, 'N' (number of participants analyzed) signifies the number of participants analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 443
percentage of participants
  None | 66.5
  Relapse | 27.3
  Breakthrough | 6.0

12. Secondary Outcome: Percentage of Participants With Viral Relapse or Breakthrough According to Cumulative Dose of Ribavirin
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. In participants with virological response, positive HCV titers measured during 24-week follow-up was interpreted as viral relapse, and positive HCV titers measured during the treatment period was interpreted as viral breakthrough. Percentage of participants with viral relapse or breakthrough in each cumulative dose group is presented. Cumulative dose was calculated as: (administered dose divided by planned dose) multiplied by 100. Percentage of participants with no relapse/breakthrough (none), with relapse, and with breakthrough in each cumulative dose group (<60%, 60-69%, 70-79%, 80-89%, and >90%) is reported.
Time Frame: Up to 24 weeks after EOT (maximum up to 96 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 391
percentage of participants
  Cumulative dose <60%: None (n=33) | 57.58
  Cumulative dose <60%: Relapse (n=33) | 39.39
  Cumulative dose <60%: Breakthrough (n=33) | 3.03
  Cumulative dose = 60-69%: None (n=21) | 66.67
  Cumulative dose = 60-69%: Relapse (n=21) | 33.33
  Cumulative dose = 60-69%: Breakthrough (n=21) | 0.00
  Cumulative dose = 70-79%: None (n=32) | 53.13
  Cumulative dose = 70-79%: Relapse (n=32) | 40.63
  Cumulative dose = 70-79%: Breakthrough (n=32) | 6.25
  Cumulative dose = 80-89%: None (n=50) | 52.00
  Cumulative dose = 80-89%: Relapse (n=50) | 38.00
  Cumulative dose = 80-89%: Breakthrough (n=50) | 10.00
  Cumulative dose >90%: None (n=257) | 70.98
  Cumulative dose >90%: Relapse (n=257) | 23.92
  Cumulative dose >90%: Breakthrough (n=257) | 5.10
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin; The relationship between the cumulative dose of ribavirin and relapse rate was analyzed using Chi-square test; Test type: Superiority or Other; p = 0.1499, Chi-squared

13. Secondary Outcome: Percentage of Participants With Viral Relapse or Breakthrough According to Starting Dose of Ribavirin
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. In participants with virological response, positive HCV titers measured during 24-week follow-up was interpreted as viral relapse, and positive HCV titers measured during the treatment period was interpreted as viral breakthrough. Percentage of participants with no relapse/breakthrough (none), with relapse, and with breakthrough in each dose group (600 mg, 800 mg, 1000 mg, 1200 mg, and 1400 mg) is presented.
Time Frame: Week 4, 12, 24, at EOT Visit, 24 weeks after EOT (maximum up to 96 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 441
percentage of participants
  Starting dose = 600mg: None (n=2) | 100.00
  Starting dose = 600mg: Relapse (n=2) | 0.00
  Starting dose = 600mg: Breakthrough (n=2) | 0.00
  Starting dose = 800mg: None (n=25) | 80.00
  Starting dose = 800mg: Relapse (n=25) | 8.00
  Starting dose = 800mg: Breakthrough (n=25) | 12.00
  Starting dose = 1000mg: None (n=171) | 66.08
  Starting dose = 1000mg: Relapse (n=171) | 29.82
  Starting dose = 1000mg: Breakthrough (n=171) | 4.09
  Starting dose = 1200mg: None (n=217) | 66.36
  Starting dose = 1200mg: Relapse (n=217) | 27.19
  Starting dose = 1200mg: Breakthrough (n=217) | 6.45
  Starting dose = 1400mg: None (n=26) | 57.69
  Starting dose = 1400mg: Relapse (n=26) | 30.77
  Starting dose = 1400mg: Breakthrough (n=26) | 11.54
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin; The relationship between the starting dose of ribavirin and relapse rate was analyzed using Chi-square test; Test type: Superiority or Other; p = 0.5885, Chi-squared

14. Secondary Outcome: Percentage of Participants With Viral Relapse or Breakthrough According to Body Weight-normalized Dose of Ribavirin
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. In participants with virological response, positive HCV titers measured during 24-week follow-up was interpreted as viral relapse, and positive HCV titers measured during the treatment period was interpreted as viral breakthrough. Percentage of participants with no relapse/breakthrough (none), with relapse, and with breakthrough in each body weight-normalized dose group (<5mg/kg/day, 5-10 mg/kg/day, 10-15 mg/kg/day, 15-20 mg/kg/day, and >20 mg/kg/day) is presented.
Time Frame: Up to 24 weeks after EOT (maximum up to 96 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 442
percentage of participants
  Ribavirin dose <5mg/kg/day: None (n=2) | 0.00
  Ribavirin dose <5mg/kg/day: Relapse (n=2) | 100.00
  Ribavirin dose <5mg/kg/day: Breakthrough (n=2) | 0.00
  Ribavirin dose = 5-10 mg/kg/day: None (n=28) | 60.71
  Ribavirin dose = 5-10 mg/kg/day: Relapse (n=28) | 35.71
  Ribavirin dose = 5-10mg/kg/day: Breakthrough(n=28) | 3.57
  Ribavirin dose = 10-15 mg/kg/day: None (n=249) | 60.64
  Ribavirin dose = 10-15 mg/kg/day: Relapse (n=249) | 30.52
  Ribavirin dose =10-15mg/kg/day:Breakthrough(n=249) | 8.84
  Ribavirin dose = 15-20 mg/kg/day: None (n=151) | 76.82
  Ribavirin dose = 15-20 mg/kg/day: Relapse (n=151) | 20.53
  Ribavirin dose=15-20mg/kg/day: Breakthrough(n=151) | 2.65
  Ribavirin dose >20 mg/kg/day: None (n=12) | 83.33
  Ribavirin dose >20 mg/kg/day: Relapse (n=12) | 16.67
  Ribavirin dose >20 mg/kg/day: Breakthrough (n=12) | 0.00
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin; The relationship between the body weight-normalized dose of ribavirin and relapse rate was analyzed using Chi-square test; Test type: Superiority or Other; p = 0.0062, Chi-squared

15. Secondary Outcome: Percentage of Participants With Viral Relapse or Breakthrough According to Dose Reduction of Ribavirin
Description: Determination of HCV titers was performed by using the COBAS AmpliPrep/COBAS TaqMan HCV technique, upon decision of the treating physician and respecting the therapeutic protocol for the treatment of hepatitis C. In participants with virological response, positive HCV titers measured during 24-week follow-up was interpreted as viral relapse, and positive HCV titers measured during the treatment period was interpreted as viral breakthrough. Percentage of participants with no relapse/breakthrough (none), with relapse, and with breakthrough in each dose-reduction group (none, dose reduction within 12 weeks, dose reduction after 12 weeks, dose reduction not specified) is presented.
Time Frame: Up to 24 weeks after EOT (maximum up to 96 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 443
percentage of participants
  No Dose Reduction: None (n=278) | 70.00
  No Dose Reduction: Relapse (n=278) | 23.57
  No Dose Reduction: Breakthrough (n=278) | 6.43
  Within 12 weeks: None (n=87) | 57.47
  Within 12 weeks: Relapse (n=87) | 35.63
  Within 12 weeks: Breakthrough (n=87) | 6.90
  After 12 weeks: None (n=57) | 63.16
  After 12 weeks: Relapse (n=57) | 33.33
  After 12 weeks: Breakthrough (n=57) | 3.51
  Not specified: None (n=19) | 68.42
  Not specified: Relapse (n=19) | 26.32
  Not specified: Breakthrough (n=19) | 5.26

ADVERSE EVENTS:
Time Frame: 96 weeks
Description: Safety population included all participants enrolled for the study.
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 52/697
Other Adverse Events (participants affected / at risk) | 353/697
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Ribavirin (N=697)
Anaemia (Blood and lymphatic system disorders) | 14
Haemolysis (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal polyp (Gastrointestinal disorders) | 1
Unevaluable event (General disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Abdominal wall abscess (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 2
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Cutaneous sarcoidosis (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Ribavirin (N=697)
Anaemia (Blood and lymphatic system disorders) | 103
Leukopenia (Blood and lymphatic system disorders) | 39
Neutropenia (Blood and lymphatic system disorders) | 37
Thrombocytopenia (Blood and lymphatic system disorders) | 40
Asthenia (General disorders) | 51
Fatigue (General disorders) | 91
Influenza like illness (General disorders) | 65
Pyrexia (General disorders) | 49
Decreased appetite (Metabolism and nutrition disorders) | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 49
Alopecia (Skin and subcutaneous tissue disorders) | 49
Pruritus (Skin and subcutaneous tissue disorders) | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.